CLINICAL TRIAL: NCT01309048
Title: Magnetic Resonance-Guided High Intensity Focused Ultrasound for Palliation of Painful Skeletal Metastases - A Pilot Study
Brief Title: Magnetic Resonance-Guided High Intensity Focused Ultrasound for Palliation of Painful Skeletal Metastases
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Philips Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02082011
Record Dates: First submitted 2011-03-02; First posted 2011-03-04 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Bone Metastasis
Keywords: bone metastasis; Patients with bone metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with painful bone metastasis (Experimental): Patients with bone metastasis causing pain
  Interventions: Device: Philips MR-guided HIFU system

INTERVENTIONS:
Device: Philips MR-guided HIFU system — HIFU is the use of focused ultrasound energy to penetrate through soft tissue and causes localized high temperatures (55°C to 70°C) for a few seconds within the target producing well defined regions of protein and nerve denaturation, irreversible cell damage, and coagulative necrosis.
  Other Names: HIFU; Ablation; High Intensity Focused Ultrasound

SUMMARY:
This study is to confirm the safety and technical of MRI guided High Intensity Focused Ultrasound (HIFU) for Palliation for Pain of Skeletal Metastases.

MRI guided high intensity focused ultrasound uses ultrasound to heat and thermally ablate tissue. The MRI system identifies the ultrasound path and monitors heat rise in the tissue. The goal of the study is to show treatment safety and effectiveness. MR-guided HIFU will be performed in patients who pass inclusion/exclusion criteria.

DETAILED DESCRIPTION:
Bone metastases are common among patients with advanced cancer and have been reported in up to 85% of cancer patients at autopsy. Complications of bone metastases include pain, functional limitation, decreased quality of life, pathological fracture, spinal cord compression and cauda equina syndrome.

External beam radiotherapy is the current standard treatment for patients with painful uncomplicated bone metastases. Unfortunately up to 30 % of patients treated with radiotherapy do not respond to therapy, and 30% of responders have their pain recur at some point after treatment. Radiotherapy re-treatment is also limited by cumulative doses delivered to sensitive structures. Ablative techniques such as cryotherapy and percutaneous radiofrequency ablation are not similarly limited by cumulative effects, however, they are invasive procedures that place patients at risk of complications.

MR-guided high intensity focused ultrasound (MR-HIFU) is a non-invasive, outpatient modality being investigated for the treatment of cancer. In MR-HIFU, a specially designed transducer is used to focus a beam of ultrasound energy into a small volume at a specific target site in the body. The focused beam produces therapeutic hyperthermia in the target field but only harmlessly warms the immediately surrounding tissue. Magnetic resonance (MR) imaging is used both to focus the ultrasound beam on the target field in the bone (the metastatic lesion and adjacent periosteum containing the nerves and vasculature for the tumor) and to perform real-time thermal mapping at and around the target. The mechanism of action of pain response is thought to be thermal periosteal denervation and / or thermal ablation of the tumor mass that diminishes pressure on the surrounding tissue.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Able to give informed consent
* Weight <140kg
* Radiologic evidence of bone metastases from any solid tumor
* Able to characterize pain specifically at the site of interest (target lesion)
* Pain score related to target lesion of ≥4 on a 0-10 point scale irrespective of medications
* Target lesion accessible for MR-HIFU procedure
* Target lesion maximum dimension ≤8cm
* Target lesion is uncomplicated (i.e.: no fracture / spinal cord compression / cauda equina syndrome / soft tissue component)
* Target lesion visible by non-contrast MRI
* Interface between bone and skin lies ≥1cm from surface
* Able to communicate sensation during MR-HIFU treatment
* MR-HIFU treatment date ≥2 weeks from most recent treatment of primary tumor or any chemotherapy.

Exclusion Criteria:

* Prior radiotherapy / surgery / ablative therapy / other local therapy to target lesion.
* Unable to characterize pain specifically at the site of interest (target lesion)
* Pregnant / Nursing woman
* Target lesion is complicated (i.e.: presence of one of fracture / spinal cord compression / cauda equina syndrome / soft tissue component).
* Target lesion <1cm from nerve bundles / bladder / bowel
* Target lesion in contact with hollow viscera
* Target lesion located in skull, spine (excluding sacrum which is allowed) or sternum
* Scar along proposed HIFU beam path
* Orthopaedic implant along proposed HIFU beam path or at site of target lesion.
* Serious cardiovascular, neurological, renal or hematological chronic disease
* Active infection
* Unable to tolerate required stationary position during treatment
* Allergy to MRI contrast agent or sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Reduction of Pain Score | 90 Days
  Determine the efficacy of MR-Guided HIFU in reducing pain scores related to the site treated as measured on the Brief Pain Inventory (BPI).
Reduction of Pain Medication | 90 Days
  Determine the efficacy of MR-Guided HIFU in reducing pain medication usage
Complications and Adverse Events | 90 Days
  Document complications and adverse events as well as the number of unintended lesions that occur as a result of treatment with MR-Guided HIFU.

SECONDARY OUTCOMES:
Changes in bone density | 90 Days
  Measure changes in bone density between X-ray and CT images taken prior to and following treatment.
Quality of Life | 90 Days
  Measure patient quality of life using both the EORTC QLQ-BM22 and FACT-BP scales

CONTACTS AND LOCATIONS:
Overall Officials: Greg Czarnota, M.D., Principal Investigator — Radiation Oncology, Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Chow E, Wu JS, Hoskin P, Coia LR, Bentzen SM, Blitzer PH. International consensus on palliative radiotherapy endpoints for future clinical trials in bone metastases. Radiother Oncol. 2002 Sep;64(3):275-80. doi: 10.1016/s0167-8140(02)00170-6. PMID 12242115